CLINICAL TRIAL: NCT06811298
Title: The Effect of Breast Massage and Virtual Reality Application on Lactation in Postpartum Women: A Randomized Controlled Trial
Brief Title: The Effect of Breast Massage and Virtual Reality Application on Lactation in Postpartum Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Şeyma Çatalgöl, Dr, Uşak University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 478-478--25
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Lactation; Lactation Disorder - Postpartum Condition or Complication; Lactation Disorder With Baby Delivered
Keywords: lactation; lactation disorder-postpartum condition or complication; lactation disorder with baby delivered
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Breast Massage (Experimental): In the breast massage group, a breast massage will be applied for 15 minutes.
- Virtual Reality (Experimental): The virtual reality group's participants will be shown a 15-minute virtual reality video depicting a river and a forest, with the aim of creating a relaxing and calming environment.
  Interventions: Other: Virtual Reality
- Control Group (No Intervention): No intervention will be applied.

INTERVENTIONS:
Other: Breast massage — The breast massage group will receive a 15-minute breast massage administered by the researchers at postoperative Day 0, Hour 3, and Hour 24. The aim of this intervention is to increase lactation. Following the interventions, mothers will be asked to breastfeed their infants, and the infants will be weighed both before and after breastfeeding.
Other: Virtual Reality — Postpartum women who undergo virtual reality headset application will watch a 15-minute river and forest video using the headset on postoperative day 0, hour 3, and hour 24. This intervention aims to help them feel in a relaxing and soothing environment and to increase lactation. Following the interventions, mothers will be asked to breastfeed their infants, and the infants will be weighed both before and after breastfeeding.
  Arms: Virtual Reality

SUMMARY:
This randomized controlled study aims to examine the effects of breast massage and virtual reality applications on breastfeeding in women after cesarean delivery. The study will include mothers aged 18-45, who have delivered a healthy baby via cesarean section at an Obstetrics and Gynecology Department of a University Training and Research Hospital located in the Aegean Region. Participants will have no health issues preventing breastfeeding, will have previously received breastfeeding counseling, and will be included after providing informed consent following the explanation of the study's objectives.

The primary research questions addressed in this study are as follows: Does breast massage applied to women after cesarean delivery affect breastfeeding? Does the application of virtual reality to women after cesarean delivery affect breastfeeding?

The research groups will be randomly assigned into three groups-virtual reality, breast massage, and control-before any interventions are applied. Randomization will be performed using the website www.randomizer.org to determine the group allocation for each participant.

In this study, 31 mothers in the virtual reality group will be shown a 15-minute virtual reality video, depicting a river and forest, viewed through a virtual reality headset, in order to create a relaxing and calming environment. This will be done on post-operative day 0, at the 3rd hour, and at the 24th hour. In the breast massage group, 32 mothers will receive breast massage for 15 minutes, administered by the researchers at the same time points (post-operative day 0, 3rd hour, and 24th hour). After the interventions, mothers will be asked to breastfeed their babies, and the babies will be weighed both before and after breastfeeding.

The control group will receive no intervention and will receive standard care (31 women). Infant weight measurements will also be taken at the same times in the control group. After the interventions, the LATCH Breastfeeding Charting System and Documentation Tool, along with the Breastfeeding Self-Efficacy Scale, will be applied to all groups on post-operative day 0, at the 3rd hour, and at the 24th hour.

A descriptive information form will be used to determine the sociodemographic and obstetric features of the participants in the study.

DETAILED DESCRIPTION:
Intervention with Virtual Reality:

The use of virtual reality (VR) applications in breastfeeding support after cesarean delivery represents a rare approach in which psychological relaxation is combined with physiological effects. In our study, VR facilitates the relaxation of new mothers through visual and auditory natural landscapes, while also exploring how this technology alleviates stress and anxiety during the breastfeeding process and its effects on milk production, thus filling a unique gap in the literature. Although VR has typically been used in the treatment of psychological disorders in other studies, systematically addressing its concrete effects on breastfeeding provides a new perspective.

The Role of Post-Cesarean Breast Massage in Early Lactation:

The enhancement of lactation after cesarean delivery is generally limited to breastfeeding counseling and psychological support. However, breast massage, as a direct physiological intervention, may play an important role in overcoming physiological barriers caused by cesarean delivery. Given the limited number of studies examining the mechanisms through which breast massage increases milk production, investigating its early-stage effects, particularly in supporting lactation after cesarean delivery, offers an innovative contribution.

Multidimensional and Comprehensive Evaluation Methods:

Rather than using a single measurement tool, our study will combine different scales, such as the LATCH Breastfeeding Charting System and the Postnatal Breastfeeding Self-Efficacy Scale, and will evaluate lactation by weighing the babies before and after the interventions. This multidimensional approach will assess not only milk production and breastfeeding success but also critical factors such as the mother's self-confidence and emotional state. This comprehensive data collection allows for a deeper understanding not only of the effectiveness of individual interventions but also of mothers' overall experiences during the breastfeeding process.

Personalized Intervention Approach:

In our research, the interventions and follow-up processes applied to each group reflect a personalized approach. Both virtual reality and breast massage will help individuals relax and breastfeed more effectively, while the control group will only undergo milk production tracking. This provides a solid foundation for comparing the effectiveness of these two methods. Moreover, highlighting the differences between the groups will contribute to the development of tailored care strategies for mothers who have undergone cesarean delivery.

These unique elements will not only contribute to the existing literature but will also bring a new perspective to clinical applications. The combination of virtual reality and physical massage offers an innovative approach that can provide valuable and unique findings related to the post-cesarean breastfeeding process.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-45 years
* Singleton pregnancy in the current gestation
* Having received breastfeeding counseling during the current pregnancy
* Gestational age between the 38th and 42nd week
* Newborn birth weight between 2500-4000 grams
* No requirement for intensive care for either the mother or the newborn

Exclusion Criteria:

* Multiple pregnancy in the current gestation
* Any mental or physical health issues that would prevent breastfeeding
* Uterine atony
* Use of medications that would require stopping breastfeeding
* Any condition that interferes with breastfeeding
* Congenital anomalies in the newborn (such as cleft palate or cleft lip) that could affect breastfeeding
* Requirement for intensive care for either the newborn or the mother

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 94 (Actual)
Dates: Start 2025-01-31 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
The amount of milk produced during breastfeeding | Post op 24 hour
  After the interventions (post-operative day 0, at the 3rd hour, and at the 24th ), mothers will be asked to breastfeed their babies, and the babies will be weighed both before and after breastfeeding.
Breastfeeding self-efficacy assessment | Post op 24 hour
  After the interventions along with the Breastfeeding Self-Efficacy Scale, will be applied to all groups on post-operative day 0, at the 3rd hour, and at the 24th hour. The Breastfeeding Self-Efficacy Scale (Dennis and Faux, 1999) is a 33-item scale developed to assess how confident mothers feel about breastfeeding. All items in the scale have positive connotations. As a result of internal consistency analysis, items with a total-item correlation below 0.60 were removed, and a 14-item short form was created. The Cronbach's alpha value for this short form is 0.94. The scale is a 5-point Likert type, with scores ranging from 14 to 70, and a higher score indicates greater breastfeeding self-efficacy. The Turkish adaptation was carried out by Aluş-Tokat and Okumuş (2010), and the Cronbach's alpha value was found to be 0.86.
Breastfeeding evaluation | Post op 24 hour
  After the interventions, the LATCH Breastfeeding Charting System and Documentation Tool, will be applied to all groups on post-operative day 0, at the 3rd hour, and at the 24th hour. The LATCH Breastfeeding Diagnostic Tool, developed in 1986, is a tool created by adapting the APGAR score system in terms of its scoring method. This measurement tool was developed to make an objective diagnosis of breastfeeding, identify breastfeeding problems, create an educational plan, establish a common language among healthcare professionals, and be used in research (to determine breastfeeding success in longitudinal studies). The tool consists of five evaluation criteria, and the first letters of these criteria combine to form the acronym LATCH. Each item is evaluated between 0-2 points. The maximum score that can be obtained from the scale is 10. In Turkey, its reliability was studied by Yenal and Okumuş (2003), and and the Cronbach's alpha value was determined to be 0.95.

CONTACTS AND LOCATIONS:
Overall Officials: Şeyma Çatalgöl, Dr, Principal Investigator — Uşak University
Locations (1):
- Uşak University, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No